CLINICAL TRIAL: NCT03308513
Title: Determination of Risk Factors and Mortality for Pediatric Chronic Critical Illnes in Turkey: Multicenter Study
Brief Title: Determination of Risk Factors and Mortality for Pediatric Chronic Critical Illness in Turkey
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other); Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hilmi Demirkiran, MD, Assistant Professor, Yuzuncu Yil University
Other Study IDs: Pediatric critical illness
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Critical Illness
Keywords: Prolonged acute mechanical ventilation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is predicted that the number of Pediatric Chronic Critical Illness increases similar to adult all over the world. The prevalence of Pediatric Chronic Critical Illness in Turkey is unknown. The investigators aimed to evaluate the etiology, comorbid conditions, demographic data, prevalence, mortality and costs of these patient in intensive care units in Turkey. In this multi-centered study, The investigators will retrospectively review the last 3 year of patients receiving treatment at the Intensive Care Unit.

DETAILED DESCRIPTION:
Patients receiving acute critical cause of ICU in the Intensive Care Unit (ICU) may be hospitalized for longer periods of time due to accompanying diseases or iatrogenic causes. This disease is called "Chronic Critical Illness" (CCI). CCI is associated with prolonged acute mechanical ventilation, but there is no definition in the literature for newborns. Pediatric CCI is estimated to be similar to adults. In the United States, the number of CCI is around 250,000, which is estimated to have doubled in the last 10 years. 50% of patients die in one year and much less than 12% recover. The estimated annual cost for the CCI in the United States is over $ 20 billion. The prevalence of Pediatric CCI in Turkey is unknown. In this study, it was aimed to investigate risk factors, mortality and cost of children with chronic critically ill and newborn patients in intensive care units in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Critical IIlness
* The patients who are younger than 18 years old and staying in ICU for at least 14 days.

(The patients who is newborn and stay in the intensive care unit for 30 days in addition to prematurity).

At least one of the additional criteria;

* Prolonged acute mechanical ventilation
* Tracheostomy
* Sepsis
* Severe wound (burn) or trauma
* Encephalopathy (Post resuscitation syndrome, Asphyxia, Intra-cranial hemorrhage, Metabolic disease, etc.)
* Traumatic brain injury
* Status epilepticus
* Post operative (Cardiac and noncardiac)
* Neuromuscular disease (Spinal Muscular Dystrophy, Cerebral Palsy, Muscular Dystrophy)

Exclusion Criteria:

* Patients with a disease other than a chronic critical disease
* Patients older than 18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are younger than 18 years or are in intensive care unit
Sampling Method: Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Critical care unit mortality | 30 Day, 90 Day, 180 Day, 365 day
  The mortality change rates in the 30th Day, 90th Day, 180th Day, 365th Day

SECONDARY OUTCOMES:
Critical care unit costs for infant patients | Duration of intensive care unit stay (From 14 day to 1 years after hospitalization)
  Cost of patients staying in intensive care unit
Critical care unit costs for premature newborn | Duration of intensive care unit stay (From 1 month to 1 year after hospitalization)
  Cost of patients staying in intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Hilmi Demirkiran, Asist.prof., Principal Investigator — Department of Anethesiology and Reanimation
Locations (1):
- Yuzuncu Yil University, School of Medicine, Van, Tusba / Zeve Kampus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demirkiran H, Kilic M, Tomak Y, Dalkiran T, Yurttutan S, Basaranoglu M, Tuncer O, Derme T, Tekeli AE, Bahar I, Keskin S, Oksuz H. Evaluation of the incidence, characteristics, and outcomes of pediatric chronic critical illness. PLoS One. 2021 May 28;16(5):e0248883. doi: 10.1371/journal.pone.0248883. eCollection 2021. PMID 34048449